CLINICAL TRIAL: NCT02203513
Title: A Phase II Single Arm Pilot Study of the Chk1/2 Inhibitor (LY2606368) In BRCA1/2 Mutation Associated Breast or Ovarian Cancer, Triple Negative Breast Cancer, and High Grade Serous Ovarian Cancer
Brief Title: A Phase II Single Arm Pilot Study of the Chk1/2 Inhibitor (LY2606368) in BRCA1/2 Mutation Associated Breast or Ovarian Cancer, Triple Negative Breast Cancer, High Grade Serous Ovarian Cancer, and Metastatic Castrate-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Eli Lilly prematurely terminated the study.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jung-Min Lee, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140156; 14-C-0156
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Results first posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer; Breast Cancer; Prostate Cancer
Keywords: p53 Dysfunction; Cell Cycle Arrest; Checkpoint Kinases; DNA Damage Repair Pathways; Hereditary Breast and Ovarian Cancer Syndrome
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome | interventions — prexasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1-Prexasertib (Experimental): Prexasertib (LY2606368) monotherapy treatment
  Interventions: Drug: LY2606368

INTERVENTIONS:
Drug: LY2606368 — 105 mg/m^2 intravenous (IV) once every 14 days of a 28 day cycle
  Other Names: Prexasertib

SUMMARY:
Background:

* All cells go through cycles which allow them to divide. In normal cells, checkpoint kinase 1 (Chk1) and checkpoint kinase 2 (Chk2) (CHEK 2 (Chk1/2) stop cell division at various points to allow any damage to deoxyribonucleic acid (DNA) to be repaired.
* When Chk1/2 are not present, cells stop dividing and eventually die. Chk1/2 Inhibitor (Prexasertib (LY2606368) blocks the Chk1/2 proteins.
* Researchers hope that by blocking Chk1/2, it will cause tumor cells to die, thereby shrinking tumors.

Objective:

- To see if LY2606368 helps shrink tumors in patients with certain breast, ovarian or prostate cancers.

Eligibility:

- Participants at least 18 years old with breast or ovarian cancer. They must have a mutation in BRCA1 BReast CAncer gene 1 and BRCA2 BReast CAncer gene 2 (BRCA1/2) genes for group 1, high grade serious ovarian cancer without BRCA1/2 mutation for group 2, or triple negative breast cancer without BRCA1/2 mutation for group 3, or prostate cancer with or without BRCA1/2 mutation for group 4.

Design:

* Participants will be screened with a medical history and physical exam. They will have blood tests, an electrocardiogram (ECG) heart test, scans, and X-rays. They will have a piece of their tumor removed at entry (computed tomography (CT)-assisted biopsy).
* Study Day 1: Participants will have a physical exam and blood drawn. They may have a CT scan of the chest, abdomen, and pelvis.
* Day 1 and Day 15 of each 28-day cycle: Participants will receive the study drug through an intravenous (IV).
* Vital signs will be checked before and after. An ECG will be done within 1 hour after.
* Day 15 and Day 28: Participants will have a physical exam, blood drawn, and a 12 lead ECG.
* Cycle 1: Participants will have weekly phone calls and blood draws. Participants may have another CT-assisted biopsy at the end of cycle 1.
* Cycle 2 and beyond, blood will be drawn every other week for routine blood tests.
* Participants will have an after-study visit with a physical exam and blood tests. Participants may have another biopsy when they progressed on treatment. They will have scans of the chest, pelvis, and abdomen and a 12 lead ECG.

DETAILED DESCRIPTION:
Background:

* Checkpoint kinases 1 and 2 (Chk1/2) are major regulators of the cell cycle and are intimately associated with the cellular response to deoxyribonucleic acid (DNA) damage and repair. Chk1/2 also function as the primary mediators of cell cycle arrest in tumors with tumor protein P53 (p53) dysfunction, such as high-grade serous ovarian cancer (HGSOC), and triple negative breast cancer (TNBC).
* Participants with germline BRCA1 BReast CAncer gene 1 and BRCA2 BReast CAncer gene 2 (BRCA1/2) mutation have inherent defects in DNA damage repair pathways.
* Chk1/2 inhibition alone yielded DNA damage and mitotic catastrophe preclinically, even in the absence of DNA damage by external agents in tumors with underlying DNA repair dysfunction.
* The second-generation Chk1/2 inhibitor (Prexasertib (LY2606368) yielded safety and preliminary single agent activity in advanced cancer participants.
* We hypothesize that LY2606368 will result in clinical benefit in participants with Germline BRCA-Mutated (gBRCAm)-associated breast or ovarian cancers, and HGSOC and TNBC with low genetic risk.

Objectives:

* To determine the objective response rate (Complete Response (CR)+Partial Response (PR) of single agent LY2606368 in patients with gBRCAm-associated breast or ovarian cancer, HGSOC and TNBC with low genetic risk.
* To determine the safety and toxicity, and progression-free interval (PFI) of LY2606368 in pretreated participants.
* To determine biochemical changes in the DNA damage repair and cell cycle check point pathways in tumor and blood samples in response to treatment.
* To determine potential resistance mechanisms to LY2606368 treatment in HGSOC.

Eligibility:

* Participants with recurrent/refractory BReast CAncer gene (BRCA) mutant breast or ovarian cancer, HGSOC, and TNBC, for whom there remains no standard curative measures.
* A documented deleterious germline or somatic BRCA mutation for breast or ovarian cancer participants enrolling in Cohort 1.
* Negative BRCA mutation testing or negative family history of hereditary breast and ovarian cancer syndrome for HGSOC (Cohort 2).
* Negative BRCA mutation testing or negative family history of hereditary breast and ovarian cancer syndrome for TNBC (Cohort 3).
* Effective with amendment I (version date 4/24/2017), Metastatic Castration-Resistant Prostate Cancer (mCRPC), Cohort 4 was closed.
* Negative BRCA mutation testing or negative family history of hereditary breast and ovarian cancer syndrome for recurrent platinum-resistant HGSOC with measurable and biopsiable disease (Cohort 5).
* Negative BRCA mutation testing or negative family history of hereditary breast and ovarian cancer syndrome for recurrent platinum-resistant HGSOC with measurable but without biopsiable disease (Cohort 6).
* Participants must be off prior chemotherapy, radiation therapy, hormonal therapy, or biological therapy for at least 4 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 and adequate organ and marrow function.

Design:

* This is an open label, single arm phase II trial to examine activity of LY2606368 in participants in the 6 independent cohorts (Cohorts 1-6).
* LY2606368 will be dosed at the recommended phase 2 dose (RP2D) of 105 mg/m^2 intravenous (IV) once every 14 days of a 28 day-cycle.
* Research samples including whole blood, circulating tumor cells (CTCs), and tumor biopsies will be obtained for pharmacodynamics (PD) endpoints at baseline, Cycle 1 Day 15 (6-24hour (hr) post-2nd dose), and/or at progression in all participants. Tumor biopsies will not be performed in Cohort 6.
* Participants (Cohorts 1-3, 5 and 6) will be evaluated every two cycles for response using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and every cycle for safety using Common Terminology Criteria for Adverse Events (CTCAE) v4.0.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. A documented deleterious germline breast cancer 1 and breast cancer 2 mutation (gBRCA1/2m) obtained in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory, including but not limited to Myriad Genetics, either by multi-gene panels or individual testing, for Cohort 1 participants prior to study enrollment. Participants with documented somatic BReast CAncer gene (BRCA) mutation obtained in a CLIA-certified laboratory also will be considered for Cohort 1. Variants of uncertain significance (VUS) of BRCA1/2 are not considered deleterious. Participants with variant of uncertain significance (VUS) or deleterious mutation in other genes without gBRCA1/2m can be considered for Cohort 2 or 3 or 5.
  2. Participants enrolling in the sporadic high grade serous epithelial or high grade endometrioid ovarian cancer group, Cohort 2, must have a negative family history of hereditary breast ovarian cancer (HBOC) syndrome, or negative gBRCA1/2m mutation test.
  3. Participants enrolling in the triple negative breast cancer (estrogen receptor (ER)-/progesterone receptor (PR)-/human epidermal growth factor receptor 2 (Her2)-) group, Cohort 3, must have a negative family history of HBOC syndrome, or negative gBRCA1/2m test. A family history of HBOC is defined by National Comprehensive Cancer Network® (NCCN®) Genetic/Familial High-Risk Assessment: Breast and Ovarian guideline.
  4. For Cohorts 1-3, 5 and 6: participants must have breast and/or epithelial or endometrioid ovarian cancer, primary peritoneal cancer, and/or fallopian tube cancer histologically or cytologically confirmed at the National Cancer Institute (NCI) that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective. ER/PR/HER2 status needs to be documented either by an outside source or at NCI. Participants with gBRCA1/2m with history of or active breast and ovarian cancers are considered for Cohort 1.

     Participants enrolling in Cohort 5, the recurrent platinum-resistant sporadic high grade serous epithelial or high grade endometrioid ovarian cancer group, must have a negative family history of HBOC syndrome, or negative gBRCA1/2m test. Participants should have recurrent platinum-resistant - defined as disease recurrence by imaging within 6 months of the last receipt of platinum-based chemotherapy. Rising mucin 16 (CA125) only is not considered as platinum-resistant disease. Participants with primary platinum refractory disease defined as progression during or within 3 months after receiving first-line platinum-based chemotherapy are not eligible.
  5. All participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral computed tomography (CT) scan.
  6. All participants except Cohort 6 must have at least one lesion deemed safe to biopsy and be willing to undergo a mandatory baseline biopsy. For Cohort 5, the second biopsy at progression is mandatory for the responders (Partial Response (PR)/Complete Response (CR)/Stable Disease (SD) > 4 months.
  7. Participants enrolling in Cohort 6, the recurrent platinum-resistant sporadic high grade serous epithelial or high grade endometrioid ovarian cancer group, must have a negative family history of HBOC syndrome, or negative gBRCA1/2m test. Participants should have recurrent platinum-resistant, defined as disease recurrence by imaging within 6 months of the last receipt of platinum-based chemotherapy. This cohort should have measurable (defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1) but without biopsiable disease, determined by principal investigator (PI) and Interventional Radiology (e.g., cystic abnormal mass, not safely biopsiable disease). Rising CA125 only is not considered as platinum-resistant disease. Participants with primary platinum refractory disease defined as progression during or within 3 months after receiving first-line platinum-based chemotherapy are not eligible.
  8. Participants must be at least 4 weeks from previous therapy (chemotherapy, hormonal therapy, and radiation therapy, or investigational agents; 6 weeks for mitomycin C).
  9. The use of raloxifene, denosumab, or bisphosphonates for bone health is allowed.
  10. There is no limit on the number of prior therapies.
  11. Participants must be at least 1 week from the last dose of complementary or alternative medications.
  12. Participants who have had major surgery must be fully recovered and greater than or equal to 4 weeks postoperative prior to enrolling on study.
  13. Age greater than or equal to 18 years.
  14. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
  15. Participants must have normal organ and marrow function (in the absence of transfusion 24 hours prior to dosing) as defined below:

      leukocytes greater than or equal to 3,000/mcL

      absolute neutrophil count greater than or equal to 1,500/mcL

      platelets greater than or equal to 100,000/mcL

      hemoglobin greater than or equal to 10mg/dL

      total bilirubin less than or equal to 1.5 X institutional upper limit of normal

      Aspartate aminotransferase (AST) Serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase (SGPT) less than or equal to 3 X institutional upper limit of normal

      creatinine less than or equal to 1.5 X institutional upper limit of normal

      OR

      measured creatinine clearance greater than or equal to 45 mL/min/1.73 m^2 for participants with

      creatinine levels above institutional normal.
  16. Potassium (K) should be within the range of greater than or equal to 3.6 mEq/L.
  17. Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to the start of the study.
  18. The effects of Chk1/2 Inhibitor (Prexasertib LY2606368) on the developing human fetus are unknown. For this reason, all subjects of reproductive potential must agree to use adequate contraception prior to study entry, for the duration of study participation, and for at least four months following the last dose of experimental therapy. All subjects of reproductive potential must also agree to use both a barrier method and a second method of birth control during the course of the study and for four months after the last dose of study drug(s). Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
  19. Ability of subject to understand, adhere to protocol requirements and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Participants who are receiving any other investigational agents.
2. Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with brain metastases diagnosed greater than 1 year prior to study entry may be considered if they received sterilizing therapy to the central nervous system (CNS) (resection or radiation) and have been CNS recurrence-free for the 1-year period.
3. Participants who have had prior treatment with LY2606368 or other Chk inhibitors
4. Participants with a serious cardiac condition, such as congestive heart failure; New York Heart Association Class III/IV heart disease; unstable angina pectoris; myocardial infarction within the last 3 months; valvulopathy that is severe, moderate, or deemed clinically significant despite medical intervention; or arrhythmias that are symptomatic or refractory to medical intervention.
5. Participants who have corrected QT interval (QTc) interval of > 470 msec on a screening electrocardiogram.
6. Participants with a prior history of drug-induced serotonin syndrome, or a family history of long-QT syndrome.
7. Lack of recovery of prior adverse events due to prior cancer therapy to Grade less than or equal to 1 (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE); except alopecia). Electrolyte abnormalities that are corrected with supplementation will be eligible. Participants with platinum-related grade 2 or greater hypomagnesemia (on replacement) will be eligible. Stable persistent grade 2 peripheral neuropathy may be allowed as determined on a case-by-case basis at the discretion of the principal investigator (PI).
8. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, clinically significant gastrointestinal (GI) bleeding or hemoptysis within 28 days prior to the start of the study, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Participants with active infection will not be eligible but may become eligible once infection has resolved and they are at least 7 days from completion of antibiotics.
10. Another previous or current invasive malignancy within the last 2 years, with the exception of curatively treated stage IA cervical carcinoma, or resected stage IA endometrial cancer, and noninvasive nonmelanoma skin cancers. Participants with gBRCA1/2m and primary breast or ovarian cancers will be eligible for Cohort 1.
11. Human immunodeficiency virus (HIV)-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with LY2606368. HIV- positive participants who are not on highly active antiretroviral therapy (HAART) and have cluster of differentiation 4 (CD4) counts > 500 will be considered on an individual basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Min Lee, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
For All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
  In addition, all large-scale genomic sequencing data will be shared with subscribers to database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol genomic data sharing plan (GDS) for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).
  Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Jin T, Xu L, Wang P, Hu X, Zhang R, Wu Z, Du W, Kan W, Li K, Wang C, Zhou Y, Li J, Liu T. Discovery and Development of a Potent, Selective, and Orally Bioavailable CHK1 Inhibitor Candidate: 5-((4-((3-Amino-3-methylbutyl)amino)-5-(trifluoromethyl)pyrimidin-2-yl)amino)picolinonitrile. J Med Chem. 2021 Oct 28;64(20):15069-15090. doi: 10.1021/acs.jmedchem.1c00994. Epub 2021 Oct 19. PMID 34665631
- [Derived] Lee JM, Nair J, Zimmer A, Lipkowitz S, Annunziata CM, Merino MJ, Swisher EM, Harrell MI, Trepel JB, Lee MJ, Bagheri MH, Botesteanu DA, Steinberg SM, Minasian L, Ekwede I, Kohn EC. Prexasertib, a cell cycle checkpoint kinase 1 and 2 inhibitor, in BRCA wild-type recurrent high-grade serous ovarian cancer: a first-in-class proof-of-concept phase 2 study. Lancet Oncol. 2018 Feb;19(2):207-215. doi: 10.1016/S1470-2045(18)30009-3. Epub 2018 Jan 18. PMID 29361470
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0156.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohorts 5 & 6 are combined because they are for platinum resistant BRCA wild type high grade serous ovarian cancer (HGSOC) participants, literally the same population. Only difference between the two cohorts is cohort 5 is a research biopsy cohort & cohort 6 had no safely biopsiable disease. Given that Eli Lilly prematurely terminated the study we could not enroll enough number of participants for both cohorts. Thus, it is appropriate and scientifically relevant to report the data in one group.
Groups:
- Cohort 1 Breast/Ovarian Breast Cancer (BRCA) Mutation Positive: All participants received Prexasertib (LY2606368) 105 mg/m^2 on dose level 1.
- Cohort 2 Breast/Ovarian Breast Cancer (BRCA) Wild-Type (wt) Cohort: All participants received Prexasertib (LY2606368) 105 mg/m^2 on dose level 1, except six participants who received Prexasertib 105 mg/m^2 on dose level 1 followed by 80 mg/m^2 on dose level -1. And one participant did not receive drug.
- Cohort 3 Breast Cancer (BRCA) Wild-Type (wt) Triple Negative Breast Cancer: All participants received Prexasertib (LY2606368) 105 mg/m^2 on dose level 1, except two participants who received Prexasertib 105 mg/m^2 on dose level 1 followed by 80 mg/m^2 on dose level -1.
- Cohort 4 Castration-resistant Metastatic Prostate: One participant received Prexasertib (LY2606368) 105 mg/m^2 on dose level -1 followed by Prexasertib 80 mg/m^2 on dose level -1. And one participant received Prexasertib 105 mg/m^2 on dose level 1.
- Cohorts 5 and 6 Ovarian Breast Cancer (BRCA) Wild-Type (wt) Platinum-resistant: All participants received Prexasertib (LY2606368) 105 mg/m^2 on dose level 1, except six participants in cohort 5 received Prexasertib 105 mg/m^2 on dose level 1 followed by 80 mg/m^2 on dose level -1. And three participants on cohort 6 received Prexasertib 105 mg/m^2 on dose level 1 followed by 80 mg/m^2 on dose level -1.
Period: Overall Study
Arm/Group | Cohort 1 Breast/Ovarian Breast Cancer (BRCA) Mutation Positive | Cohort 2 Breast/Ovarian Breast Cancer (BRCA) Wild-Type (wt) Cohort | Cohort 3 Breast Cancer (BRCA) Wild-Type (wt) Triple Negative Breast Cancer | Cohort 4 Castration-resistant Metastatic Prostate | Cohorts 5 and 6 Ovarian Breast Cancer (BRCA) Wild-Type (wt) Platinum-resistant
Started | 22 | 29 | 9 | 2 | 49
Completed | 16 | 21 | 6 | 1 | 43
Not Completed | 6 | 8 | 3 | 1 | 6
Not completed — Refused further treatment | 2 | 0 | 1 | 0 | 0
Not completed — Switched to alternative treatment | 3 | 4 | 0 | 0 | 4
Not completed — Did not receive investigational product (IP) | 0 | 1 | 0 | 0 | 0
Not completed — Death (unrelated to study therapy) | 1 | 3 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Cohorts 5 & 6 are combined because they are for platinum resistant BRCA wild type high grade serous ovarian cancer (HGSOC) participants, literally the same population. Only difference between the two cohorts is cohort 5 is a research biopsy cohort & cohort 6 had no safely biopsiable disease. Given that Eli Lilly prematurely terminated the study we could not enroll enough number of participants for both cohorts. Thus, it is appropriate and scientifically relevant to report the data in one group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Breast/Ovarian Breast Cancer (BRCA) Mutation Positive | Cohort 2 Breast/Ovarian Breast Cancer (BRCA) Wild-Type (wt) Cohort | Cohort 3 Breast Cancer (BRCA) Wild-Type (wt) Triple Negative Breast Cancer | Cohort 4 Castration-resistant Metastatic Prostate | Cohorts 5 and 6 Ovarian Breast Cancer (BRCA) Wild-Type (wt) Platinum-resistant | Total
Number analyzed (Participants) | 22 | 29 | 9 | 2 | 49 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 6 | 1 | 26 | 64
  >=65 years | 6 | 14 | 3 | 1 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.32 (9.55) | 64.61 (9.52) | 52.46 (15.17) | 65.6 (10.04) | 62.59 (10.84) | 61.31 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 9 | 0 | 49 | 109
  Male | 0 | 0 | 0 | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 21 | 28 | 9 | 2 | 47 | 107
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 5 | 1 | 4 | 11
  White | 20 | 27 | 4 | 1 | 42 | 94
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 29 | 9 | 2 | 49 | 111

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete Response (CR) + Partial Response (PR)
Description: Objective response (CR+PR) of single agent Prexasertib (LY2606368) in participants with germline BReast CAncer gene -Mutated (gBRCAm)-associated breast and ovarian cancers, high grade serous ovarian cancer (HGSOC) and triple-negative breast cancer (TNBC) at low genetic risk. Response was measured using the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Complete Response is disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Cohorts 1-3, 5, & 6 were restaged every 2 mos. Cohort 4 was restaged every 3 mos. Restaging continued until participant's disease was deemed progressive by RECIST or until removed from treatment for other etiology for an combined average of 133 days.
Population: Overall, 17 participants were not evaluable for this outcome measure. Overall participants analyzed adjusted to include only evaluable subjects as defined by the protocol (i.e., only those participants who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated; Response Evaluation Criteria in Solid Tumors (RECIST) Evaluable).
Measure: Count of Participants; unit: Participants
Groups:
- Cohorts 5 and 6 Ovarian Breast Cancer (BRCA) Wild-Type (wt) Platinum-resistant: Cohorts 5 and 6 are combined because they are for platinum resistant BRCA wild type high grade serous ovarian cancer (HGSOC) participants, literally the same population. Only difference between the two cohorts is cohort 5 is a research biopsy cohort and cohort 6 had no safely biopsiable disease. Given that Eli Lilly prematurely terminated the study we could not enroll enough number of participants for both cohorts.
  All participants received Prexasertib (LY2606368) 105 mg/m^2 on dose level 1, except six participants in cohort 5 received Prexasertib 105 mg/m^2 on dose level 1 followed by 80 mg/m^2 on dose level -1. And three participants on cohort 6 received Prexasertib 105 mg/m^2 on dose level 1 followed by 80 mg/m^2 on dose level -1.
Arm/Group | Cohort 1 Breast/Ovarian Breast Cancer (BRCA) Mutation Positive | Cohort 2 Breast/Ovarian Breast Cancer (BRCA) Wild-Type (wt) Cohort | Cohort 3 Breast Cancer (BRCA) Wild-Type (wt) Triple Negative Breast Cancer | Cohort 4 Castration-resistant Metastatic Prostate | Cohorts 5 and 6 Ovarian Breast Cancer (BRCA) Wild-Type (wt) Platinum-resistant
Number analyzed (Participants) | 20 | 26 | 8 | 1 | 39
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 2 | 8 | 1 | 0 | 12

2. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Participants were followed for the duration of treatment and up to 4 weeks after being off treatment, an average of 7 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Cohorts 5 and 6 Breast Cancer (BRCA) Wild-Type (wt) Platinum Resistant Cohort: All participants received Prexasertib (LY2606368) 105 mg/m^2 on dose level 1, except four participants in cohort 5 received Prexasertib 105 mg/m^2 on dose level 1 followed by 80 mg/m^2 on dose level -1. And one participant on cohort 6 received Prexasertib 105 mg/m^2 on dose level 1 followed by 80 mg/m^2 on dose level -1.
Arm/Group | Cohort 1 Breast/Ovarian Breast Cancer (BRCA) Mutation Positive | Cohort 2 Breast/Ovarian Breast Cancer (BRCA) Wild-Type (wt) Cohort | Cohort 3 Breast Cancer (BRCA) Wild-Type (wt) Triple Negative Breast Cancer | Cohorts 5 and 6 Ovarian Breast Cancer (BRCA) Wild-Type (wt) Platinum-resistant | Cohorts 5 and 6 Breast Cancer (BRCA) Wild-Type (wt) Platinum Resistant Cohort
Number analyzed (Participants) | 22 | 29 | 9 | 2 | 49
Participants | 22 | 29 | 9 | 2 | 49

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of treatment and up to 4 weeks after being off treatment, an average of 7 months.
Description: Cohorts 5 & 6 are combined because they are for platinum resistant BRCA wild type high grade serous ovarian cancer (HGSOC) participants, literally the same population. Only difference between the two cohorts is cohort 5 is a research biopsy cohort &cohort 6 had no safely biopsiable disease. Given that Eli Lilly prematurely terminated the study we could not enroll enough number of participants for both cohorts. Thus, it is appropriate and scientifically relevant to report the data in one group.
Arm/Group | Cohort 1 Breast/Ovarian Breast Cancer (BRCA) Mutation Positive | Cohort 2 Breast/Ovarian Breast Cancer (BRCA) Wild-Type (wt) Cohort | Cohort 3 Breast Cancer (BRCA) Wild-Type (wt) Triple Negative Breast Cancer | Cohort 4 Castration-resistant Metastatic Prostate | Cohorts 5 and 6 Ovarian Breast Cancer (BRCA) Wild-Type (wt) Platinum-resistant
All-Cause Mortality (participants affected / at risk) | 1/22 | 3/29 | 1/9 | 0/2 | 2/49
Serious Adverse Events (participants affected / at risk) | 10/22 | 12/29 | 3/9 | 1/2 | 28/49
Other Adverse Events (participants affected / at risk) | 22/22 | 29/29 | 9/9 | 2/2 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Breast/Ovarian Breast Cancer (BRCA) Mutation Positive (N=22) | Cohort 2 Breast/Ovarian Breast Cancer (BRCA) Wild-Type (wt) Cohort (N=29) | Cohort 3 Breast Cancer (BRCA) Wild-Type (wt) Triple Negative Breast Cancer (N=9) | Cohort 4 Castration-resistant Metastatic Prostate (N=2) | Cohorts 5 and 6 Ovarian Breast Cancer (BRCA) Wild-Type (wt) Platinum-resistant (N=49)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (5) | 0 (0) | 1 (1) | 4 (5)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 7 (9)
Fever (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 7 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Paralysis of lower extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Death from progressive disease (PD)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PD (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 3 (5)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Breast/Ovarian Breast Cancer (BRCA) Mutation Positive (N=22) | Cohort 2 Breast/Ovarian Breast Cancer (BRCA) Wild-Type (wt) Cohort (N=29) | Cohort 3 Breast Cancer (BRCA) Wild-Type (wt) Triple Negative Breast Cancer (N=9) | Cohort 4 Castration-resistant Metastatic Prostate (N=2) | Cohorts 5 and 6 Ovarian Breast Cancer (BRCA) Wild-Type (wt) Platinum-resistant (N=49)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 9 (12) | 13 (19) | 2 (2) | 1 (1) | 23 (40)
Activated partial thromboplastin time prolonged (Investigations) | 6 (16) | 15 (33) | 6 (8) | 1 (1) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (9) | 6 (7) | 0 (0) | 0 (0) | 13 (16)
Alkaline phosphatase increased (Investigations) | 9 (12) | 11 (26) | 0 (0) | 1 (1) | 19 (26)
Allergic reaction (Immune system disorders) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 22 (81) | 26 (158) | 9 (39) | 2 (2) | 44 (256)
Anorexia (Metabolism and nutrition disorders) | 7 (9) | 8 (9) | 2 (2) | 2 (2) | 16 (17)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 4 (11) | 5 (40) | 0 (0) | 0 (0) | 6 (10)
Aspartate aminotransferase increased (Investigations) | 7 (12) | 5 (7) | 1 (1) | 0 (0) | 10 (17)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (12) | 6 (7) | 1 (1) | 1 (1) | 14 (21)
Bloating (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 7 (10)
Blood and lymphatic system disorders - Other, Petechia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 8 (9)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 4 (4)
Chills (General disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (13) | 9 (12) | 0 (0) | 1 (2) | 14 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8) | 2 (2) | 0 (0) | 9 (9)
Creatinine increased (Investigations) | 7 (10) | 11 (30) | 1 (1) | 1 (1) | 15 (27)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (6)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 14 (24) | 4 (5) | 2 (2) | 26 (46)
Dizziness (Nervous system disorders) | 3 (4) | 4 (4) | 0 (0) | 0 (0) | 8 (11)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (11) | 3 (4) | 0 (0) | 15 (22)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (2) | 4 (4) | 1 (1) | 1 (1) | 12 (15)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Eye infection (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, Eye ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, Infection (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 10 (21) | 19 (29) | 6 (7) | 1 (1) | 39 (72)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 9 (17) | 9 (13) | 3 (3) | 0 (0) | 13 (24)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 8 (10)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 7 (7)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 6 (7)
Gastrointestinal disorders - Other, Early satiety (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Mouth Sore (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Mouth ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 6 (11)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (8)
Hemorrhoids (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 4 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 6 (8) | 0 (0) | 0 (0) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (13) | 9 (33) | 2 (3) | 1 (1) | 13 (25)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (3) | 3 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6) | 5 (8) | 1 (3) | 1 (1) | 10 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (10) | 6 (15) | 2 (6) | 1 (1) | 22 (64)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5) | 11 (17) | 1 (1) | 0 (0) | 7 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 4 (6)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (8)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Thrush (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Viral origin-shingles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 8 (8)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 17 (85) | 26 (159) | 8 (37) | 1 (1) | 41 (205)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8)
Malaise (General disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Right lower extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, lower extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 11 (15) | 20 (27) | 3 (5) | 2 (2) | 28 (47)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 4 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Fluid from mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Thyroid adenomatoid nodule, R lobe
Nervous system disorders - Other, Cauda Equina Syndrome 2/2 bone lesions (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, L chin weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 19 (59) | 27 (138) | 8 (27) | 1 (4) | 44 (99)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 3 (4) | 0 (0) | 0 (0) | 6 (9)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Pain (General disorders) | 4 (5) | 4 (5) | 0 (0) | 1 (1) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 7 (8)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 17 (74) | 24 (168) | 9 (29) | 1 (1) | 46 (244)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3) | 1 (2) | 0 (0) | 8 (10)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (7) | 1 (1) | 0 (0) | 1 (1) | 6 (6)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Nitrite positive urine (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 5 (9) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Abrasion of LUE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Eccchymosis on forearm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Herpes zoster (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, oral blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 3 (6) | 2 (2) | 1 (1) | 0 (0) | 2 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (7) | 1 (1) | 0 (0) | 8 (9)
Surgical and medical procedures - Other, Biliary stent placed (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (1) | 5 (7) | 0 (0) | 0 (0) | 5 (7)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (7) | 2 (2) | 0 (0) | 14 (29)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (6) | 13 (21) | 0 (0) | 1 (1) | 13 (26)
Vulval infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 10 (13)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 19 (76) | 28 (179) | 9 (35) | 1 (2) | 44 (47)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT02203513/Prot_SAP_000.pdf
  • Informed Consent Form: Standard Consent (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT02203513/ICF_001.pdf
  • Informed Consent Form: Cohort: All Participants Consent (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT02203513/ICF_002.pdf